CLINICAL TRIAL: NCT00402493
Title: A Prospective,Randomized,Masked,Study to Evaluate the Interaction of Non-Steroidal Anti-Inflammatory Agent With IOP-Lowering Effect of Brimonidine or Latanoprost.
Brief Title: Study to Determine if Taking OTC Non-Steroidal Anti-Inflammatory Affects Eye Pressure in Patients Using Glaucoma Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philadelphia Eye Associates (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GA6110HV
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2017-09

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular Hypertension; Xalatan; Alpahgan; Ibuprofen; Non-Steroidal Anti-Inflammatory; Brimonidine; Latanoprost; Eye Pressure; Intra-Ocular Pressure
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Ibuprofen; Latanoprost; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Latanoprost (Active Comparator): to determine whether commonly used OTC non-steroidal anti-inflammatory agents taken orally has any effect on the ability of either latanoprost or brimonidine to lower high eye pressure
  Interventions: Drug: ibuprofen, latanoprost, brimonidine; Drug: Ibuprofen, brimonidine, latanoprost
- Brimonidine (Active Comparator): to determine whether commonly used OTC non-steroidal anti-inflammatory agents taken orally has any effect on the ability of either latanoprost or brimonidine to lower high eye pressure
  Interventions: Drug: ibuprofen, latanoprost, brimonidine; Drug: Ibuprofen, brimonidine, latanoprost
- ibuprofen (Active Comparator): to determine whether commonly used OTC non-steroidal anti-inflammatory agents taken orally has any effect on the ability of either latanoprost or brimonidine to lower high eye pressure
  Interventions: Drug: ibuprofen, latanoprost, brimonidine; Drug: Ibuprofen

INTERVENTIONS:
Drug: ibuprofen, latanoprost, brimonidine — to determine whether commonly used OTC non-steroidal anti-inflammatory agents taken orally has any effect on the ability of either latanoprost or brimonidine to lower high eye pressure
  Other Names: placebo
Drug: Ibuprofen, brimonidine, latanoprost — to determine whether commonly used OTC non-steroidal anti-inflammatory agentsn(200mg ibuprofen) taken orally has any effect on the ability of either latanoprost or brimonidine to lower high eye pressure
  Other Names: ibuprofen 200mg, and placebo pills
  Arms: Brimonidine; Latanoprost
Drug: Ibuprofen — ibuprofen 200mg
  Other Names: ibuprofen 200mg
  Arms: ibuprofen

SUMMARY:
The Purpose of This Study is to Determine if Taking an Over the Counter Non-Steroidal Anti-Inflammatory(Ibuprofen)has an Effect on Eye Pressure in Patients using Brimonidine(Alphagan)and Latanoprost(Xalatan) eye drops.

DETAILED DESCRIPTION:
Topical IOP-lowering therapy has the advantage of providing a drug level directly to the end organ with very little or no systemic absorption thereby reducing side effect potential. There is very little information in the ophthalmic literature regarding potential drug interactions between topical IOP-lowering medications and other medications taken orally for other medical reasons. Patients will be randomized to either latanoprost or brimonidine. Patients in both groups will be randomized to either placebo or ibuprofen for the first 14 days and then crossed over to the other treatment for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral or unilateral primary open angle glaucoma or ocular hypertension
* An IOP in each eye of greater than 22mm HG after washout of IOP lowering medications
* No worse than 20/200 best corrected visual acuity
* Normal appearing or non-occludable anterior chamber angles
* Discontinuation of current POAG or OH medications before participation in the study.
* Written Informed Consent

Exclusion Criteria:

* Use of any other ocular medications
* Previous ocular surgery or laser therapy within the last three months.
* Systemic treatment with any adrenergic agonist or antagonist, corticosteroid or nonsteroidal anti-inflammatory agents(low dose apsirin will be accepted if dose remains the same for entire study period).
* An age of less than 21,of child bearing age and currently pregnant, considering pregnancy or a nursing mother.
* A history of medical noncompliance or unreliability.
* Presence of uncontrolled hypertension, cardiac arrhythmia, cerebrovascular accident, nasal polyps, bleeding diathesis, peptic ulcer disease, gastritis or known intolerance, contraindication or allergy to any drugs used in the study.
* Lactose Intolerance.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph I. Markoff, Ph.D,M.D, Principal Investigator — Philadelphia Eye Associates
Locations (2):
- United States (2):
  - Philadelphia Eye Associates, Willingboro, New Jersey
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania